CLINICAL TRIAL: NCT05833256
Title: Inflammation-related Markers for the Prediction of Postoperative 1-year Mortality in Patients Undergoing Valvular Heart Surgery
Brief Title: A Prediction Model for 1-year Mortality After Valvular Heart Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-1117
Record Dates: First submitted 2023-02-28; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Patients Undergoing Valvular Heart Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to develop a predictive model for mortality incorporating nutritional, inflammatory, and perioperative factors in patients undergoing valvular heart surgery. In this retrospective study, the investigators aimed to establish a comprehensive prediction model to predict the risk of 1-year mortality in valvular heart surgery patients through the identification of the inflammatory index most associated with 1-year mortality and developing a prognostic nomogram model incorporating perioperative risk factors with nutritional and inflammatory indices that would be verified by validation cohorts.

ELIGIBILITY:
Inclusion Criteria:

1) patients who presented for surgery primarily due to valvular heart disease, including those who required concomitant coronary artery bypass surgery, aortic procedures, or other cardiac procedures.

Exclusion Criteria:

1. patients aged <18 years
2. undergoing transcatheter valve replacement, combined congenital heart surgery, or implantation of ventricular assist device, 3) lacking data required for calculating inflammatory indices, or 4) follow-up loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care hospital
Sampling Method: Probability Sample
Enrollment: 2046 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
1-year mortality after valvular heart surgery | 1 year after valvular heart surgery
  Mortality at follow-up was analysed using time-to-event analysis, with survival time defined as the time from date of surgery until date of death.

SECONDARY OUTCOMES:
neutrophil-to-lymphocyte ratio (NLR), calculated as the number of neutrophils divided by the number of lymphocytes | within 1 month before surgery
  the white blood cell count with (neutrophil)
monocyte-to-lymphocyte ratio (MLR), calculated as the number of monocytes divided by the number of lymphocytes | within 1 month before surgery
  the white blood cell count with ( monocyte)
platelet-to-lymphocyte ratio (PLR), calculated as the number of platelets divided by the number of lymphocytes | within 1 month before surgery
  the white blood cell count with platelet

CONTACTS AND LOCATIONS:
Overall Officials: Jin Sun Cho, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No